CLINICAL TRIAL: NCT05378165
Title: Three Distraction Methods for Pain Reduction During Colonoscopy: A Randomized Controlled Trial Evaluating the Effects on Pain and Anxiety
Brief Title: Three Distraction Methods for Pain Reduction During Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Selda Karaveli Çakır, Assistant professor, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020-KAEK-143-146
Record Dates: First submitted 2022-04-29; First posted 2022-05-18 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Colonoscopy; Colon Disease
Keywords: pain; anxiety; music; stress ball; virtual reality; nursing
MeSH Terms: conditions — Colonic Diseases; Pain; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Single centre, open-label, randomized, parallel-group trial
Who Masked: Outcomes Assessor
Masking Description: While participants and researchers were not blinded to group allocation, the biostatistician remained blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Music group (Experimental): The music group listened to Acemasiran-type classical Turkish music with a headset from an MP3 player starting at about 10 min before colonoscopy until completion of the procedure.
  Interventions: Other: Music group
- Stress ball group (Experimental): The stress ball group was given stress balls which was medium hard and made of high-quality silicone approximately 10 minutes before colonoscopy. The patients in stress ball group were instructed to "squeeze the balls twice after counting up to five" and "repeat until the end of the entire procedure".
  Interventions: Other: Stress ball group
- Video group (Experimental): The patients in the video group allowed to watch a licensed virtual reality application, "A walk on the beach", through an Android mobile phone placed in Cardboard Super Flex Goggles, started 10 minute before the colonoscopy until the procedure was completed.
  Interventions: Other: Video group
- Control group (Other): Standard colonoscopy was performed on the patients in the control group, without any additional intervention.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Music group — The study was divided into three stages; before; during; and after colonoscopy. Patient's hemodynamics parameters, including systolic and diastolic blood pressures, heart rate, and oxygen saturation, were measured about 5 to 10 min before, during and within 10 min after the colonoscopy procedure was complete. All of the patients who participated in the study underwent the standard protocol used in the Endoscopy Unit of our institution. Colonoscopy was performed on patients in all groups without the use of anesthesia. After positioning the patients in the left lateral position for the colonoscopy procedure, and vemcain local anesthetic and vaseline was applied to the anal area before starting colonoscopy using a Fujinon flexible colonoscope. The music group listened to Acemasiran-type classical Turkish music.Acemasiran-type music affects the human brain and provides a sense of creativity to people. This musical tone has pain- relieving and antispasmodic
  Arms: Music group
Other: Stress ball group — The study was divided into three stages; before; during; and after colonoscopy. Patient's hemodynamics parameters, including systolic and diastolic blood pressures, heart rate, and oxygen saturation, were measured about 5 to 10 min before, during and within 10 min after the colonoscopy procedure was complete. Colonoscopy was performed on patients in all groups without the use of anesthesia. After positioning the patients in the left lateral position for the colonoscopy procedure, and vemcain local anesthetic and vaseline was applied to the anal area before starting colonoscopy using a Fujinon flexible colonoscope. The stress ball group was given stress balls which was medium hard and made of high-quality silicone approximately 10 minutes before colonoscopy. The patients in stress ball group were instructed to "squeeze the balls twice after counting up to five" and "repeat until the end of the entire procedure".
  Arms: Stress ball group
Other: Video group — The study was divided into three stages; before; during; and after colonoscopy. Patient's hemodynamics parameters, including systolic and diastolic blood pressures, heart rate, and oxygen saturation, were measured about 5 to 10 min before, during and within 10 min after the colonoscopy procedure was complete.
  All of the patients who participated in the study underwent the standard protocol used in the Endoscopy Unit of our institution. Colonoscopy was performed on patients in al groups without the use of anesthesia. After positioning the patients in the left lateral position for the colonoscopy procedure, and vemcain local anesthetic and vaseline was applied to the anal area before starting colonoscopy using a Fujinon flexible colonoscope. Video group allowed to watch a licensed virtual reality application,"A walk on the beach", through an Android mobile phone placed in Cardboard Super Flex Goggles, started 10 minute before the colonoscopy until the procedure was completed.
  Arms: Video group
Other: Control group — The study was divided into three stages; (1) before; (2) during; and (3) after colonoscopy. Patient's hemodynamics parameters, including systolic and diastolic blood pressures, heart rate, and oxygen saturation, were measured about 5 to 10 min before, during and within 10 min after the colonoscopy procedure was complete.
  All of the patients who participated in the study underwent the standard protocol used in the Endoscopy Unit of our institution. Colonoscopy was performed on patients in al groups without the use of anesthesia. After positioning the patients in the left lateral position for the colonoscopy procedure, and vemcain local anesthetic and vaseline was applied to the anal area before starting colonoscopy using a Fujinon flexible colonoscope. Control group, without any additional intervention.
  Arms: Control group

SUMMARY:
Colonoscopy is a common procedure to evaluate the gastrointestinal tract. The colonoscopy procedure can sometimes be uncomfortable and painful for the patient.

The aim of this study was to compare the effects on pain and anxiety of distraction methods used during colonoscopy. Single centre, randomized, parallel-group trial.

Endoscopy unit of a training and research hospital in northern Turkey A total of 120 patients were recruited and randomized into four groups as music, stress ball, video, and control group. The data were collected using Visual Analog Scale for pain and satisfaction, State-Trait Anxiety Inventory for anxiety, and hemodynamic parameters.

Data collection continues

DETAILED DESCRIPTION:
Colonoscopy is one of the endoscopic procedures used for the diagnostic and interventional procedures of the intestines. Compared to other radiological imaging methods, the most important advantage of colonoscopy is that it can be used to evaluate symptoms and complaints as well as to obtain a biopsy when a differential diagnosis is needed. In recent years, therefore, colonoscopy has been recognized as the gold standard for colon cancer screening. Most patients consider colonoscopy a painful and uncomfortable procedure. Studies revealed that patients experience moderate anxiety during the colonoscopy procedure. The reflex spasm resulting from stimulation of the colon in order to obtain a better image during colonoscopy, and acute distension resulting from flatulence may cause patients to experience pain during and after the procedure. Studies have shown that patients experience pain and anxiety during the colonoscopy procedure. The pain and anxiety that patients experience is not only related to the procedure, but also to the stress of the likelihood of getting cancer over time. Performing colonoscopy under sedation is widely used in clinical practice. However, sedation increases complications associated with colonoscopy, and has potential risks, such as hypoxemia, hypoventilation, aspiration pneumonia, pulmonary embolism and myocardial infarction. Different drug regimens are used to manage pain during colonoscopy; however, the optimal regime is still debated. In recent years, in addition to pharmacological methods, non-pharmacological methods such as distraction applications such as music and virtual reality have been used to reduce anxiety and pain during the colonoscopy procedure.There are randomized controlled studies showing that simple distraction methods used during the colonoscopy procedure reduce pain and anxiety.Although there are few studies comparing the effectiveness of multiple simple distraction methods such as music, stress ball, and video on pain and anxiety during painful procedures, there are no studies in the literature comparing the effects of three different distraction methods during the colonoscopy procedure. The study was divided into three stages; (1) before; (2) during; and (3) after colonoscopy. Patient's hemodynamics parameters, including systolic and diastolic blood pressures, heart rate, and oxygen saturation, were measured about 5 to 10 min before, during and within 10 min after the colonoscopy procedure was complete.

All of the patients who participated in the study underwent the standard protocol used in the Endoscopy Unit of our institution. Colonoscopy was performed on patients in al groups without the use of anesthesia. After positioning the patients in the left lateral position for the colonoscopy procedure, and vemcain local anesthetic and vaseline was applied to the anal area before starting colonoscopy using a Fujinon flexible colonoscope. The patients who met the inclusion criteria were assigned to one of four groups: (1) music; (2) stress ball; (3) video or (4) control group. The patients who met the inclusion criteria were assigned to one of four groups: (1) music; (2) stress ball; (3) video or (4) control group.

The music group listened to Acemasiran-type classical Turkish music with a headset from an MP3 player starting at about 10 min before colonoscopy until completion of the procedure. Acemasiran-type music affects the human brain and provides a sense of creativity to people. This musical tone has pain- relieving and antispasmodic The stress ball group was given stress balls which was medium hard and made of high-quality silicone approximately 10 minutes before colonoscopy. The patients in stress ball group were instructed to "squeeze the balls twice after counting up to five" and "repeat until the end of the entire procedure". The patients in the video group allowed to watch a licensed virtual reality application, "A walk on the beach", through an Android mobile phone placed in Cardboard Super Flex Goggles, started 10 minute before the colonoscopy until the procedure was completed. Standard colonoscopy was performed on the patients in the control group, without any additional intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent colonoscopy without anesthesia
* Patients who were over 18 years of age
* Patients who did not have vision problems
* Patients who did not have hearing problems
* Patients who did not have cognitive problems

Exclusion Criteria:

* Patients who underwent colonoscopy with anesthesia
* Patients who were under 18 years of age
* Patients who have vision problems
* Patients who have hearing problems
* Patients who have cognitive problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Before Colonoscopy 1 | 5 to 20 min before colonoscopy
  When the patient comes to the endoscopy unit State anxiety levels (measured The State Anxiety Inventory) The State Anxiety Inventory requires individuals to described heir feelings at a specific moment under specific circumstances. Scores on the entire scale range from 20 to 80, with higher scores indicating higher anxiety levels.
Before Colonoscopy 2 | 5 to 20 min before colonoscopy
  When the patient comes to the endoscopy unit Patient's systolic blood pressure (mmHg)
Before Colonoscopy 3 | 5 to 20 min before colonoscopy
  When the patient comes to the endoscopy unit Diastolic blood pressures (mmHg)
Before Colonoscopy 4 | 5 to 20 min before colonoscopy
  When the patient comes to the endoscopy unit Heart rate (per minute)
Before Colonoscopy 5 | 5 to 20 min before colonoscopy
  When the patient comes to the endoscopy unit Oxygen saturation (SpO2)
Before Colonoscopy 6 | 5 to 20 min before colonoscopy
  When the patient comes to the endoscopy unit Pain levels (measured The Visual Analog Scale)
During colonoscopy 1 | During colonoscopy
  Patien's systolic blood pressures (mmHg) (within 5 minutes of the colonoscopy procedure)
During colonoscopy 2 | During colonoscopy
  Patient's diastolic blood pressures(mmHg) (within 5 minutes of the colonoscopy procedure)
During colonoscopy 3 | During colonoscopy
  Patient's heart rate (per minute) (within 5 minutes of the colonoscopy procedure)
During colonoscopy 4 | During colonoscopy
  Oxygen saturation (within 5 minutes of the colonoscopy procedure)
During colonoscopy 5 | During colonoscopy
  Pain were measured (measured The Visual Analog Scale) (within 5 minutes of the colonoscopy procedure) Pain intensity is scored between 0-10, absence of pain is "0" point, whereas the most severe pain is scored "10"

SECONDARY OUTCOMES:
After colonoscopy 1 | 10-15 min after the colonoscopy procedure was complete.
  Patient systolic blood pressures (mmHg) (10 minutes after colonoscopy)
After colonoscopy 2 | 10-15 min after the colonoscopy procedure was complete.
  diastolic blood pressures(mmHg) (10 minutes after colonoscopy)
After colonoscopy 3 | 10-15 min after the colonoscopy procedure was complete.
  heart rate (per minute) (10 minutes after colonoscopy)
After colonoscopy 4 | 10-15 min after the colonoscopy procedure was complete.
  Oxygen saturation (10 minutes after colonoscopy)
After colonoscopy 5 | 10-15 min after the colonoscopy procedure was complete.
  pain were measured (measured The Visual Analog Scale) (10 minutes after colonoscopy) Pain intensity is scored between 0-10, absence of pain is "0" point, whereas the most severe pain is scored "10"
After colonoscopy 6 | 10-15 min after the colonoscopy procedure was complete.
  State anxiety levels (measured The State Anxiety Inventory) (15 minutes after colonoscopy procedure) evaluated. The State Anxiety Inventory requires individuals to described heir feelings at a specific moment under specific circumstances. Scores on the entire scale range from 20 to 80, with higher scores indicating higher anxiety levels.

CONTACTS AND LOCATIONS:
Overall Officials: Selda Karaveli Çakır, PhD, Principal Investigator — Kastamonu University
Locations (1):
- Kastamonu University, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Celebi D, Yilmaz E, Sahin ST, Baydur H. The effect of music therapy during colonoscopy on pain, anxiety and patient comfort: A randomized controlled trial. Complement Ther Clin Pract. 2020 Feb;38:101084. doi: 10.1016/j.ctcp.2019.101084. Epub 2019 Dec 23. PMID 32056820
- [Background] Hudson BF, Ogden J, Whiteley MS. Randomized controlled trial to compare the effect of simple distraction interventions on pain and anxiety experienced during conscious surgery. Eur J Pain. 2015 Nov;19(10):1447-55. doi: 10.1002/ejp.675. Epub 2015 Jan 30. PMID 25641687
- [Background] Bashiri M, Akcali D, Coskun D, Cindoruk M, Dikmen A, Cifdaloz BU. Evaluation of pain and patient satisfaction by music therapy in patients with endoscopy/colonoscopy. Turk J Gastroenterol. 2018 Sep;29(5):574-579. doi: 10.5152/tjg.2018.18200. PMID 30260780
- [Background] Sargin M, Uluer MS, Aydogan E, Hanedan B, Tepe MI, Eryilmaz MA, Ebem E, Ozmen S. Anxiety Levels in Patients Undergoing Sedation for Elective Upper Gastrointestinal Endoscopy and Colonoscopy. Med Arch. 2016 Apr;70(2):112-5. doi: 10.5455/medarh.2016.70.112-115. Epub 2016 Apr 1. PMID 27147784
- [Result] Sorkpor SK, Johnson CM, Santa Maria DM, Miao H, Moore C, Ahn H. The Effect of Music Listening on Pain in Adults Undergoing Colonoscopy: A Systematic Review and Meta-Analysis. J Perianesth Nurs. 2021 Oct;36(5):573-580.e1. doi: 10.1016/j.jopan.2020.12.012. Epub 2021 May 12. PMID 33994100
- [Result] Karaveli Cakir S, Evirgen S. The Effect of Virtual Reality on Pain and Anxiety During Colonoscopy: A Randomized Controlled Trial. Turk J Gastroenterol. 2021 May;32(5):451-457. doi: 10.5152/tjg.2021.191081. PMID 34231475